CLINICAL TRIAL: NCT03514927
Title: Translation of High-intensity Focused Ultrasound (HIFU) or Treatment of Intermediate and High-Risk Prostate Cancer
Brief Title: High-Intensity Focused Ultrasound in Treating Participants With Intermediate and High-risk Prostate Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4P-17-9; NCI-2018-00605 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 4P-17-9 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2018-04-20; First posted 2018-05-03 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Prostate Cancer Stage I AJCC V6; Prostate Cancer Stage II; Prostate Cancer Stage III
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (HIFU, radical prostatectomy) (Experimental): HIFU PHASE: Participants undergo mpMRI and CEUS pre-HIFU treatment and then CEUS post-HIFU treatment. Participants then undergo HIFU treatment over 2-2.5 hours.
  PROSTATECTOMY PHASE: Within 2-4 weeks post-HIFU treatment, participants undergo mpMRI 1-2 days prior to radical prostatectomy. On the day of surgery, participants undergo CEUS prior to radical prostatectomy.
  Interventions: Procedure: Contrast-Enhanced Ultrasound; Device: High-Intensity Focused Ultrasound; Other: Laboratory Biomarker Analysis; Procedure: Multiparametric Magnetic Resonance Imaging; Procedure: Radical Prostatectomy

INTERVENTIONS:
Procedure: Contrast-Enhanced Ultrasound — Undergo CEUS
  Other Names: CEUS
Device: High-Intensity Focused Ultrasound — Under go HIFU
  Other Names: HIFU; high-intensity focused ultrasound therapy
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Multiparametric Magnetic Resonance Imaging — Undergo mpMRI
  Other Names: Multiparametric MRI
Procedure: Radical Prostatectomy — Undergo prostatectomy
  Other Names: Prostatovesiculectomy

SUMMARY:
This phase II trial studies how well high-intensity focused ultrasound works in treating participants with intermediate and high-risk prostate cancer. High-intensity focused ultrasound uses high frequency sound waves to deliver a strong beam which may target and destroy a specific part of the prostate, while minimizing damage to surrounding structures and tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Histologic assessment of cancer kill in the post high-intensity focused ultrasound (HIFU) needle biopsy and excised treated lobe 2-4 weeks after treatment with HIFU.

II. Radiologic assessment of areas suspicious for residual cancer in the treated lobe on multiparametric magnetic resonance imaging (mpMRI) and/or contrast enhanced ultrasound (CEUS) 2-4 weeks post-HIFU (immediately prior to radical prostatectomy).

SECONDARY OBJECTIVES:

I. Assessment of differences in tumor microenvironment, specifically upregulation of the immune system, before and after HIFU treatment on both the treated and untreated lobes.

II. Assessment of HIFU parameters needed to achieve dose-escalation, in the event that such escalation is needed per our study design.

OUTLINE:

HIFU PHASE: Participants undergo mpMRI and CEUS pre-HIFU treatment and then CEUS post-HIFU treatment. Participants then undergo HIFU treatment over 2-2.5 hours.

PROSTATECTOMY PHASE: Within 2-4 weeks post-HIFU treatment, participants undergo mpMRI 1-2 days prior to radical prostatectomy. On the day of surgery, participants undergo CEUS prior to radical prostatectomy.

After completion of study treatment, participants are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Male having a diagnosis of clinically-significant prostate cancer (CsPCa) made within the past 12 months (Gleason 7-9) with no evidence of metastatic disease; all outside pathology will be re-reviewed at University of Southern California (USC) to verify diagnosis
* Patients have elected to undergo radical prostatectomy (RP) as treatment of choice and have to be a surgical candidate for RP; this determination will be made by the patient in conjunction with their treating urologist and is current standard of practice
* Standard preoperative evaluation is performed and deemed satisfactory to proceed to surgery as per their treating urologist
* Ability to understand AND willingness to sign a written informed consent
* Patients must be willing to undergo HIFU, CEUS, MRI and prostate biopsy pre-RP for research purposes

Exclusion Criteria:

* Patients may not be receiving any other investigational agents or have received any definitive prostate cancer (PCa)-specific treatment (en-bloc resection of bladder tumors [EBRT], Brachytherapy etc) prior
* Patients with known metastases would be excluded from this clinical trial
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, clinical significant cardiac arrhythmia (rate controlled atrial fibrillation allowed), or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with active autoimmune diseases or active immune suppressive therapy or inflammatory bowel disease; a low dose steroid daily administration (equivalent dexamethasone < 10mg/day) is acceptable
* Patients with rectal disease
* Patients who are unable to undergo MRI
* Patients with convincing evidence of extraprostatic extension or T4 disease on digital rectal examination (DRE)

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Mean percentage of viable clinically-significant prostate cancer (Gleason pattern 4 or 5) after high-intensity focused ultrasound (HIFU) treatment | Up to 3 months
  Determined by calculating the mean percent of viable cancer tissue remaining after HIFU using two different measurements: histologic examination of excised prostate specimen and histologic examination of post HIFU needle biopsy. Each of these two measurements will be investigated independently using two types of analyses as follows: percent viable cancer in excised prostate specimen and percent viable cells using post-HIFU needle biopsy. Will calculate the mean percent viable cancer across patients along with a corresponding 95% confidence interval based on all 32 fully evaluable patients.

SECONDARY OUTCOMES:
Mean detection level of immunological factors | Up to 3 months
  Determined by immunohistochemistry (IHC) and real-time polymerase chain reaction (RT-PCR). For this will use data collected from IHC on a panel of markers, obtained from both biopsy specimens obtained in the non-treated lobe at the time of biopsy (pre-HIFU) and right before RP (post-HIFU) revisiting them same pre-HIFU biopsy sites. Will compare mean IHC levels of each antibody examined in the pre-HIFU contralateral biopsy to the post-HIFU biopsy obtained from the same site. Mean IHC levels for each antibody will be compared using exact tests and analysis of variance.

CONTACTS AND LOCATIONS:
Overall Officials: Inderbir Gill, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States